CLINICAL TRIAL: NCT01489631
Title: Comparison of Intra-articular Infiltration and Gabapentin With Epidural Analgesia After Total Knee Replacement Surgery
Brief Title: Analgesia After Total Knee Replacement Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: St. Antonius Hospital (Other)
Responsible Party: Principal Investigator, Leon Timmerman, anesthesiologist, St. Antonius Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: TKP-37796
Record Dates: First submitted 2011-12-08; First posted 2011-12-09 (Estimated); Last update posted 2015-06-08 (Estimated); Status verified 2015-06

CONDITIONS: Total Knee Arthroplasty
Keywords: Epidural; Local infiltration; Knee; Arthroplasty
MeSH Terms: interventions — Ropivacaine; Bupivacaine; Sufentanil; Gabapentin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- epidural analgesia (Active Comparator): The first group will be treated with epidural analgesia. Before surgery the epidural catheter will be placed according to local guidelines. After the operation epidural infiltration with bupivacaine and sufentanil will be commenced.
  Interventions: Drug: marcaine; Drug: sufentanil
- local infiltration (Active Comparator): The second group will receive local infiltration with ropivacaine of the knee during surgery.
  Interventions: Drug: naropin
- local infiltration and gabapentin (Active Comparator): The third group will receive local infiltration with ropivacaine of the knee during surgery and will additionally be treated with gabapentin.
  Interventions: Drug: naropin; Drug: neurontin

INTERVENTIONS:
Drug: naropin — ropivacaine 0,2%, 3x 50 ml during surgery
  Other Names: ropivacaine
  Arms: local infiltration; local infiltration and gabapentin
Drug: marcaine — bupivacaine 0,125%
  Other Names: bupivacaine
  Arms: epidural analgesia
Drug: sufentanil — sufentanil 1mcg/ml
  Other Names: sufenta forte
  Arms: epidural analgesia
Drug: neurontin — gabapentin 600 mg pre-operative 3 dd 300 mg
  Other Names: gabapentin
  Arms: local infiltration and gabapentin

SUMMARY:
Postoperative pain after total knee replacement surgery is difficult to treat. Mobilisation and hospital discharge might be delayed. Recent research shows that intra-articular infiltration with local anesthetics and perioperative prescription of gabapentin can improve outcome.

Objective of the study: Comparison of mobilisation speed and postoperative NRS-scores of patients after total knee replacement surgery which is treated with epidural analgesia or peroperative infiltration of the knee. Appraisal of the value of gabapentin for reduction of postoperative opiate consumption.

DETAILED DESCRIPTION:
Study design:

Prospective randomised study

Study population:

Patients aged eighteen years or older, in whom knee replacement surgery is indicated. They will have spinal anaesthesia and epidural analgesia if indicated by randomisation. They must not have contraindications for epidural analgesia or the used medication in this study.

Intervention:

The first group will be treated with epidural analgesia. Before surgery the epidural catheter will be placed according to local guidelines. After the operation epidural infiltration with bupivacaine and sufentanil will be commenced. The second group will receive local infiltration with ropivacaine of the knee during surgery. Half of these patients will additionally be treated with gabapentin.

Primary study parameters/outcome of the study:

NRS-score (11-scale Numeric Rating Scale in which 0 means no pain, and 10 means most pain imaginable) in rest.

Secondary study parameters/outcome of the study:

Speed of mobilisation, postoperative opiate consumption. NRS scores during flexion exercise of the knee and during walking exercise.

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older and legally responsible
* Waiting for total knee replacement surgery
* Informed consent

Exclusion Criteria:

* Contraindications for epidural analgesia
* Aortic Valve stenosis
* Severely compromised cardiac function
* infection near epidural punction site
* Redo knee surgery
* Previous arthrotomies
* Allergy/Hypersensitivity for study mediation or all other used medication
* Participation in other studies

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 81 (Actual)
Dates: Start 2013-03; Primary Completion 2014-04 (Actual); Study Completion 2014-04 (Actual)

PRIMARY OUTCOMES:
NRS score in rest | 3 days after surgery

SECONDARY OUTCOMES:
Speed of mobilisation | 3 days after surgery
Postoperative morphine consumption | 3 days after surgery
  Daily morphine consumption (mg) per day
NRS score during flexion exercise | 3 days after surgery
NRS score during walking exercise | 3 days after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Leon Timmerman, MD, Principal Investigator — Anesthesiologist; Louis N Marting, MD, Principal Investigator — Orthopedic surgeon
Locations (1):
- St. Antonius Hospital, Nieuwegein, Netherlands